CLINICAL TRIAL: NCT01675531
Title: A Multicenter, Phase IV, Interventional Study to Assess the Efficacy and Safety of Oxycodone/Naloxone in Korean Patients With Chemotherapy-Induced Peripheral Neuropathy Who Need Opioid Combination Treatment With Existing Pregabalin Treatment
Brief Title: A Study to Assess the Efficacy and Safety of Oxycodone/Naloxone in Korean Patients With Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Korea Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OXN12-KR-402
Record Dates: First submitted 2012-08-27; First posted 2012-08-30 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-10

CONDITIONS: Cancer
Keywords: Targin; Chemotherapy Induced Peripheral Neuropathy (CIPN)
MeSH Terms: conditions — Neoplasms | interventions — Oxycodone; Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Targin (Experimental): Targin
  Interventions: Drug: Targin

INTERVENTIONS:
Drug: Targin — Single arm for Targin
  Other Names: Oxycodone and Naloxone

SUMMARY:
A multicenter, phase IV, interventional study to assess the efficacy and safety of Targin (Oxycodone/Naloxone) Korean patients with CIPN (Chemotherapy-Induced Peripheral Neuropathy) who need opioid combination treatment with existing pregabalin of last dose prior to study enrollment without changing.

The investigators will assess study objectives as below.

Primary objective

* To assess the pain reduction rate after 4 weeks treatment from baseline (week 0)

Secondary objectives

* To assess the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACIT-GOG/NTX)
* To assess physician's overall satisfaction
* To assess subject's overall satisfaction
* To assess safety

The investigators have a hypothesis that Targin will show favorable efficacy & safety profile for CIPN patients.

DETAILED DESCRIPTION:
This will be a multicenter, phase IV, interventional study to assess the efficacy and safety of Targin (Oxycodone/Naloxone) Korean patients with CIPN(Chemotherapy-Induced Peripheral Neuropathy) who need opioid combination treatment with existing pregabalin of last dose prior to study enrollment without changing.

Upon providing written informed consent, subject will be screened in the study and assessment will be performed at that time such as safety data (adverse event (AE)/serious adverse events (SAEs)) including laboratory results, physical examination, vital sign, medical history taking, 24 hours pain intensity score, Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT-GOG/NTX), physician's overall satisfaction and subject's overall satisfaction. If patient is eligible in inclusion/exclusion criteria at the time of visit 1, the patient will receive treatment with Targin. Re-screening, study drug dose interruption is not allowed. The duration of study drug dose interruption is defined as for 1 week.

Treatment with Targin will be started at 10/5mg twice daily for 4 weeks, and proper titration (up-titration) will be allowed at each visit according to the investigator's decision. Dose titration up to a maximum of Targin 40/20mg twice daily will be permitted during study period.

The up-titration will be considered by investigator's judgement as followings; (1) if the rescue medication was used more than 2 times per day, on average or (2) based on the daily average Numeric Rating Scale (NRS), if the NRS was changed to worsen since the previous visit, (3) Investigator's judgement by considering any titration needed situation (e.g. dose, frequency of rescue medication).

Safety laboratories will be obtained at baseline (visit 1) and study end (visit 4) in a local laboratory. The laboratory values within 4 weeks prior to baseline (visit 1) will be allowed to use at study visit 1.

The rescue medication is the 5mg of (Immediate release codon trade mark)IRcodonTM .

Patients will be withdrawn from the study if the following circumstance require study drug discontinuation:

Failure of pain control (Failure of pain control will be decided by investigators judgement, e.g. there is poor pain control or lack of efficacy despite 2~3 times of up titration.) Adjustment of the other analgesics due to AEs except Targin or IRcodonTM Adjustment of the other major pain management modality (e.g. chemotherapy, radiotherapy, surgery, non-surgical interventional therapy, etc.) Withdrawal of informed consent Pregnancy Any other significant risk to the patient's safety in the clinical judgement of the investigator

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 20 and <80 years of age
* Patients who has diagnosed as Chemotherapy-Induced Peripheral Neuropathy by investigator's judgment
* Patient who are receiving pregabalin for the treatment of Chemotherapy- Induced Peripheral Neuropathy
* Patients who have moderate to severe pain intensity which is not controlled with 300mg of pregabalin per day for at least 1 week: NRS ≥ 4
* Patients who need opioid combination treatment with existing pregabalin treatment
* Naïve patients for strong opioid (Naïve patient defined as who did not treated for 90 days)
* Patients who signed a written informed consent form

Exclusion Criteria:

* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant. UNLESS they are:

  * women whose partners have been sterilized by vasectomy or other means
  * two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method. Adequate barrier methods of contraception include: diaphragm, condom (by the partner), intrauterine device (copper or hormonal), sponge or spermicidal. Hormonal contraceptives include any marketed contraceptive agent that includes an estrogen and/or (Progest - progesterone) progestational agent.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive urine pregnancy test
* Patients with known hypersensitivity to Oxycodone or Naloxone or to any of the excipients
* Patients with severe respiratory depression with hypoxia and/or hypercapnia
* Patients with severe chronic obstructive pulmonary disease
* Patients with cor pulmonale
* Patients with severe bronchial asthma
* Patients with non-opioid induced paralytic ileus
* Patients with moderate to severe hepatic impairment
* Targin product contains lactose. Patients with rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption should not take
* Abnormal aspartate aminotransferase (AST; SGOT), alanine aminotransferase (ALT; SGPT), or alkaline phosphatase levels (>2.5 times the upper limit of normal, it is allowed >5 times the upper limit of normal in case of transition in liver) or an abnormal total bilirubin and/or creatinine level(s) (greater than 1.5 times the upper limit of normal), gamma glutamyl transpeptidase (GGT or GGTP) ≥ 3 times the upper limit of normal
* Patients with uncontrolled seizures
* Requiring interventional treatment for pain such as neural blockade procedure or regional infusion
* Patients with increased intracranial pressure
* In the investigator's opinion, subjects who are receiving hypnotics or other central nervous system (CNS) depressants that may pose a risk of additional CNS depression with opioid study medication
* Patients with myxoedema, not adequately treated hypothyroidism or Addison's disease
* Patients receiving opioid substitution therapy for opioid addiction (e.g. methadone or buprenorphine)
* Clinically significant impairment of cardiovascular, respiratory and renal function
* Major surgery within 1 month prior to screening or planned surgery
* Chemotherapy or radiotherapy within 2 weeks prior to the screening visit, or planned chemotherapy or radiotherapy during the study period.
* Mainly pain originated other than Chemotherapy-Induced Peripheral Neuropathy
* Patients with diabetic neuropathy
* With a disability that may prevent the patient from completing all study requirements and in particular, interfere with 24hrs pain intensity score
* Patients known to have, or suspected of having a history of drug abuse
* Patients with history of opioid or drug dependence
* Any situation where opioids are contraindicated
* Having used other investigational drugs at the time of enrollment, or within 30 days of enrollment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kang, Ph.D, Principal Investigator — Seoul ST.Mary Hospital
Locations (1):
- Seoul ST.Mary Hospital, Seoul, Banpogu, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Safety set: 72 subjects ITT set: 66 subjects PP set: 41 subjects.
Pre-assignment Details: 73 Patients was enrolled. However, 1 patient was not administered investigational drug. So the patient excluded from safety set.
Groups:
- Oxycontin/Naloxone: Targin(Oxycontin/Naloxone)
  Targin: Single arm for Targin
Period: Overall Study
Arm/Group | Oxycontin/Naloxone
Started | 66
Completed | 41
Not Completed | 25
Not completed — Adverse Event | 9
Not completed — Withdrawal by Subject | 7
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 8

BASELINE CHARACTERISTICS:
Population: Safety set: 72 subjects
Groups:
- Oxycodone/Naloxone: Targin
  Targin: Single arm for Targin
Arm/Group | Oxycodone/Naloxone
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.97 (8.99)
Age, Customized [Number; unit: participants]
  18~29 | 0
  30~39 | 1
  40~49 | 4
  50~59 | 20
  60~69 | 34
  >70 | 13
Gender [Count of Participants; unit: Participants]
  Female | 21
  Male | 51

OUTCOME MEASURES:

1. Primary Outcome: NRS (Numeric Rating Scale)
Description: Change of pain intensity score via NRS after vist 4 weeks treatment from baseline (week 0).
  NRS-Pain scale assessed the severity of a subject's pain of mean pain over the past 24 hours prior to the visit on a scale of 0 (No pain) and 10 (Worst possible pain). Change = mean score at Week4/ET minus mean score at Baseline.
Time Frame: 4 weeks
Population: Analysis of ITT population set. Missing data was handled as LOCF(Last Observation Carried Forward Method).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxycodone/Naloxone
Number analyzed (Participants) | 66
units on a scale | -1.29 (1.84)

2. Secondary Outcome: Mean Change in FACT-GOG/NTX From Visit1(Week 0) to Visit 4(Week 4 Post-treatment).
Description: Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FAICT-GOG/NTX).
  The mean changes in FACT/GOG-NTX total score and each FACT/GOG-NTX subscale score from Visit 1 (Week 0) to Visit 4 (Week 4 post-treatment) were analyzed. Missing data was handled as LOCF(Last Observation Carried Forward Method).
  FACT/GOG-NTX total score range was from 0 to 152. The average change score from baseline to visit 4 indicates thay a lower score on the FACT/GOG-NTX means lower quality of life and a greater impact of neurotoxic symptom on the patient's life.
Time Frame: 4 weeks
Population: Analysis of ITT population set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxycontin/Naloxone
Number analyzed (Participants) | 66
units on a scale | -2.78 (17.66)

3. Secondary Outcome: Physician's Overall Satisfaction
Description: Physician's overall satisfaction was scored 7 scales from Very much worse to Very much improved. (Very much worse, much worse, minimally worse, No change, Minimally improved, much improved, very much improved).
Time Frame: 4 weeks
Population: Analysis of ITT population set.
Measure: Number; unit: participants
Arm/Group | Oxycontin/Naloxone
Number analyzed (Participants) | 66
participants
  Very much worse | 0
  much worse | 3
  minimally worse | 2
  No change | 25
  Minimally improved | 19
  Much improved | 16
  Very much improved | 1

4. Secondary Outcome: Patient's Overall Satisfaction
Description: Patient's overall satisfaction was assessed 7 scales from very much worse to very much improved. (Very much worse, much worse, minimally worse, no change, minimally improved, much improved, very much improved)
Time Frame: 4weeks
Population: Analysis of ITT population set.
Measure: Number; unit: participants
Arm/Group | Oxycontin/Naloxone
Number analyzed (Participants) | 66
participants
  Very much worse | 0
  Much worse | 3
  Minimally worse | 2
  No change | 26
  Minimally improved | 15
  Much improved | 18
  Very much improved | 2

ADVERSE EVENTS:
Time Frame: 4weeks
Groups:
- Oxycodone/Naloxone: Targin(Oxycodone/Naloxone)
  Targin: Single arm for Targin
Arm/Group | Oxycodone/Naloxone
Serious Adverse Events (participants affected / at risk) | 2/72
Other Adverse Events (participants affected / at risk) | 25/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone/Naloxone (N=72)
Neutrophil count decreased (Investigations) | 1 (1) — Severity was severe and causality was not suspected with investigational drug(Oxycodone/Naloxone). Action taken was not changed to dose of investigational drug. However, Eventually, patient was withdrawal to study by herself.
Mental inpairment (Nervous system disorders) | 1 (1) — Severity was mild and causality was not suspected. Action taken of study drug was not changed. The patient was completed to study by the end without drop out.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone/Naloxone (N=72)
Dizziness (Nervous system disorders) | 15 (17)
Somnolence (Nervous system disorders) | 4 (4)
Hypersomnia (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No